CLINICAL TRIAL: NCT00639483
Title: A Double-Blind, Placebo-Controlled, Randomized Study of the Efficacy of Celecoxib as Add-on Therapy to Risperidone Versus Risperidone Alone in Patients With Schizophrenia
Brief Title: Efficacy and Safety of Celecoxib as Add-on Therapy to Risperidone Versus Risperidone Alone in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COXXNT-6570-001; A3191105
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsules twice daily as add-on therapy to risperidone twice daily (range 2-8 mg/day) for 11 weeks
  Arms: A
Drug: Placebo — Matched oral placebo as add-on to risperidone twice daily (range 2-8 mg/day) for 11 weeks
  Arms: B

SUMMARY:
To assess the efficacy and safety of celecoxib as add-on therapy to risperidone versus risperidone alone in patients with schizophrenia

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of schizophrenia (according to Diagnostic and Statistical Manual of Mental Disorders [DSM]-IV-TR criteria and made by a specialist in psychiatry) and acute exacerbation of schizophrenia requiring hospitalization
* Total PANSS score of ?60 at screening
* History of schizophrenia of ?10 years (from onset of prodromal symptoms)

Exclusion criteria:

* Axis-I DSM-IV-TR diagnosis other than schizophrenia
* Less than a full cycle has lapsed at time of screening following the last injection of a depot antipsychotic
* Currently taking celecoxib or other selective cyclo-oxygenase 2 inhibitors, or other antiinflammatory medication

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2003-03; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Positive and Negative Syndrome Scale (PANSS) score | Week 11

SECONDARY OUTCOMES:
Patient-Reported Outcomes using Treatment Satisfaction Questionnaire for Medication | Week 4 and 11
Physical examination | Week 11
Laboratory exams | Weeks 1, 2, 4, 6, 8, 11
Change from baseline in Global Improvement and Efficacy Index scores of Clinical Global Impressions scale of Psychosis | Weeks 4, 6, and 11
Change from baseline in total PANSS score | Weeks 4 and 6
Change from baseline in PANSS-derived Brief Psychiatric Rating Scale score | Weeks 4, 6, and 11
Change from baseline in combined PANSS Negative plus General Psychopathology Subscale Score and the separate PANSS Psychopathology Subscale Scores | Weeks 4, 6, and 11
Change from baseline in PANSS five-factor component scores | Weeks 4, 6, and 11
Time to onset of clinically meaningful improvement in total PANSS score | Weeks 1, 2, 4, 6, 8, and 11
Adverse events | Weeks 1, 2, 4, 6, 8, 11

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Argentina (3):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Lanús, Buenos Aires
  - Pfizer Investigational Site, La Plata, Pcia. de Buenos Aires
- Brazil (5):
  - Pfizer Investigational Site, PR, Curitiba
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Aparecida de Goiânia, Goiania
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Germany (3):
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
- Pfizer Investigational Site, Mexico City, Mexico
- Philippines (2):
  - Pfizer Investigational Site, Mandaluyong
  - Pfizer Investigational Site, Pasig
- Taiwan (2):
  - Pfizer Investigational Site, Niao-Sung Hsiang, Kaohsiung
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=COXXNT-6570-001&StudyName=Efficacy%20and%20Safety%20of%20Celecoxib%20as%20Add-on%20Therapy%20to%20Risperidone%20Versus%20Risperidone%20Alone%20in%20Patients%20with%20Schizophrenia